CLINICAL TRIAL: NCT00694915
Title: Open Label, Randomized, Multicentric, Comparative and Controlled Clinical Trial to Compare the Efficacy and Toxicity of Mycobacterium w Intra-dermal to Intravesical BCG in Patients With Newly Diagnosed Superficial Transitional Cell Carcinoma With High Probability of Recurrence
Brief Title: Study of Mycobacterium w in Superficial Transitional Cell Carcinoma of Bladder
Acronym: STCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cadila Pharnmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-60/9150
Record Dates: First submitted 2008-05-29; First posted 2008-06-11 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer
Keywords: STCC (Superficial Transitional Cell Carcinoma)
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mycobacterium w vaccine; BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mw (Experimental): Mycobacterium w
  Interventions: Biological: Mycobacterium w
- BCG (Active Comparator): bacillus Calmette-Guerin (BCG)
  Interventions: Biological: BCG (Bacillus Calmette-Guerin)

INTERVENTIONS:
Biological: Mycobacterium w — Immunomodulator
  Arms: Mw
Biological: BCG (Bacillus Calmette-Guerin) — Immunotherapeutic agent
  Other Names: Bacillus Calmette Guerin
  Arms: BCG

SUMMARY:
The purpose of this study is to determine and compare the effect of this treatment on recurrence rate and to assess the toxicity in both arms of patients with STCC. Other objectives include determining the effects of this treatment on quality of life, and comparing the effect of Mycobacterium w on time to tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent.
* Patients with newly diagnosed superficial transitional cell carcinoma with completely resected papillary tumors and high probability of recurrence risk i.e. stage T1 Grade 2, T1 Grade 3 & CIS.

and Ta or T1 disease with an increased risk of recurrence defined as 2 tumors (primary and recurrent or 2 recurrences) within 1 year, 3 or more within the last 6 months and/ or carcinoma in situ on at least one random biopsy.

* 18 years or above
* ECOG of 0-2 range
* life expectancy is at least 24 weeks.
* Absolute neutrophil count≥1,500/c.mm
* platelet count≥100,000//c.mm
* Hemoglobin ≥9.0g/dL

  * No patient who has eczema will be allowed to participate in this study.
  * Patients who are immuno-compromised will not be enrolled.
  * Patients with severe hepatic dysfunctions or with evidence of Cirrhosis will not be enrolled.
  * Patients with uncontrolled diabetes mellitus will not be enrolled in the study
  * No evidence of residual tumor in the cystoscopy done 6 weeks after the TUR

Note: The effects of Investigational product on the developing human fetus is at the recommended therapeutic dose are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients who have had cytotoxic chemotherapy or radiotherapy prior to entering the study.
* No patient who has eczema should be allowed to participate in this study.
* Patients who are immuno-compromised should not be enrolled.
* Patients with severe hepatic dysfunctions or evidence of Cirrhosis should not be enrolled.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study.
* Pregnant women or nursing women are excluded from this study because agents used in the study have potential for teratogenic or abortifacient effects. Because there is known potential risk for adverse events in nursing infants secondary to treatment of the mother with investigational agent, breastfeeding should be discontinued if the mother is treated with investigational product.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Hypersensitivity to celecoxib, sulfonamides, aspirin, other NSAIDs, or any study reagent
* Previous splenectomy
* Clinically significant active infection
* Patients with uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-08-28 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
Recording of any clinical adverse reactions at anytime during the study for assessment of safety | 24 months
Recurrence Rate-Evaluated after 3 months by doing sonography, cystoscopy, and cytology | 24 months

SECONDARY OUTCOMES:
Quality of Life- The measure of an individual's sense of well-being and ability to carry out various activities | 24 months
Time to Tumor progression -will be evaluated every 3 months for 15 months during the study period | 15

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Desai, MD, Principal Investigator — Muljibhai Patel Urological Hospital; N K Mohanty, MD, Principal Investigator — V M Medical College & Safdarjang Hospital; Amillal Bhat, MD, Principal Investigator — S P Medical College & AG of Hospitals; Sujata Patwardhan, MD, Principal Investigator — Seth G S Medical College & K E M Hospital; Kim Mammen, MD, Principal Investigator — Christian Medical College, Vellore, India; Sushil Bhatia, MD, Principal Investigator — Choithram Hospital and Research Centre; B. R. Srivastav, MD, Principal Investigator — Cancer Hospital and Research Institute; Jitendra Amlani, MD, Principal Investigator — Urocare Hospital; Anup Kundu, MD, Principal Investigator — Institute of Post Graduate Medical Education & Research, S. S. K. M. Hospital; H. K. Moorthy, MD, Principal Investigator — Lourdes Hospital; Shrawan K. Singh, MD, Principal Investigator — Post Graduate Institute of Medical Education & Research; Purshottam K. Puri, MD, Principal Investigator — Indira Gandhi Medical College, Shimla; Rajeev Sood, MD, Principal Investigator — Dr. Ram Manohar Lohia Hospital & PGIMER; Padmaraj Hegde, MD, Principal Investigator — Kasturba Medical College & Hospital; Yathish Kumar, MD, Principal Investigator — N.R.R. Hospital
Locations (15):
- India (15):
  - Muljibhai Patel Urological Hospital, Nadiād, Gujarat
  - Urocare Hospital, Rajkot, Gujarat
  - Indira Gandhi Medical College, Shimla, Himachal Pradesh
  - N.R.R. Hospital, Bangalore, Karnataka
  - Kasturba Medical college and Hospital, Manipal, Karnataka
  - Lourdes Hospital, Kochi, Kerala
  - Choithram Hospital and Research Centre, Indore, Madhya Pradesh
  - Cancer Hospital and Research Institute, Gwalior, Madya Pradesh
  - Seth G S Medical College & K E M Hospital, Pārel, Mumbai
  - Christian Medical College, Ludhiana, Punjab
  - P.B.M. Hospital & A.G. of Hospitals, Bikaner, Rajasthan
  - IPGMER, S.S.K.M. Hospital, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Dr. Ram Manohar Lohia Hospital & PGIMER, New Delhi
  - V M Medical College & Safdarjang Hospital, New Delhi